CLINICAL TRIAL: NCT02287428
Title: A Phase I Study of a Personalized NeoAntigen Cancer Vaccine With Radiotherapy Plus Pembrolizumab/MK-3475 Among Newly Diagnosed Glioblastoma Patients
Brief Title: Personalized NeoAntigen Cancer Vaccine w RT Plus Pembrolizumab for Patients With Newly Diagnosed GBM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: The Ben & Catherine Ivy Foundation (Other); Accelerate Brain Cancer Cure (Other); Merck Sharp & Dohme LLC (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David Reardon, MD, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-362; 51986 (Other: Merck & Co., Inc.)
Record Dates: First submitted 2014-10-29; First posted 2014-11-10 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; pembrolizumab; Temozolomide; poly ICLC

STUDY DESIGN:
Intervention Model Description: Patients on Cohort 1 received Neovax after completing standard RT. After Cohort 1 completed accrual, we added three new cohorts (1a, 1b, & 1c); patients on Cohorts 1a, 1b, & 1c (run in parallel) receive pembrolizumab (starting at different times) in addition to standard RT + NeoVax.
Masking Description: After Cohort 1 completed accrual, new patients with MGMT-unmethylated tumors are randomized to one of three new cohorts (1a, 1b, & 1c) and new patients with MGMT-methylated tumors are registered to new cohort 1d.
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Coh 1 (Original Cohort): Standard RT Followed by NeoVax (Experimental): After the screening procedures confirm participant eligible to participate in the research study (must be registered to within 6 weeks of resection):
  * ~ 6 weeks of standard radiation therapy (RT) followed by an RT-recovery period.
  * During that time, participant NeoAntigen Vaccine-Preparation is created (process takes ~ 12 weeks)
  After participant recovers from RT and vaccine is created, participant will re-screen to confirm participant is eligible to receive study vaccinations. Once registered, participant will proceed to receive study vaccinations:
  - NeoAntigen Vaccine: NeoVax will be administered on an individual basis using a dosing schedule that incorporates both priming and boost phases (~ 7 months total: 5 priming followed by 2 boost vaccine administrations)
  Interventions: Radiation: Radiation Therapy; Biological: Personalized NeoAntigen Peptides; Biological: Poly-ICLC
- Coh 1a: Pembrolizumab w Std RT Followed by NeoVax + Pembro (Experimental): * RT: Standard RT (60Gy) over 6 weeks
  * Pembrolizumab: Starts within 2 weeks of start of RT, and continues every 3 weeks for up to 2 years
  * NeoVax: Starts in the Adjuvant setting - as soon as available after RT - and is administered on days 1, 4, 8, 15, 22 [priming doses], 78 and 134 [booster doses] o NeoVax Day 1 does not have to coincide with Pembrolizumab dosing
  Interventions: Radiation: Radiation Therapy; Biological: Personalized NeoAntigen Peptides; Drug: Pembrolizumab; Biological: Poly-ICLC
- Coh 1b: Std RT Followed by NeoVax + Pembrolizumab (Experimental): * RT: Standard RT (60Gy) over 6 weeks
  * Pembrolizumab: Starts 1-4 weeks after completion of NeoVax priming, and continues every 3 weeks for up to 2 years
  * NeoVax: Starts in the Adjuvant setting - as soon as available after RT - and is administered on days 1, 4, 8, 15, 22 [priming doses], 78 and 134 [booster doses] o NeoVax Day 1 does not have to coincide with Pembrolizumab dosing
  Interventions: Radiation: Radiation Therapy; Biological: Personalized NeoAntigen Peptides; Drug: Pembrolizumab; Biological: Poly-ICLC
- Coh 1c: Std RT (+ 1 dose Pembro) Followed by NeoVax & Pembo (Experimental): * RT: Standard RT (60Gy) over 6 weeks
  * Pembrolizumab: Single dose of pembrolizumab administered within 2 weeks of start of RT; re-starts 1-4 weeks after completion of NeoVax priming, and continues every 3 weeks for up to 2 years.
  * NeoVax: Starts in the Adjuvant setting - as soon as available after RT - and is administered on days 1, 4, 8, 15, 22 [priming doses], 78 and 134 [booster doses] o NeoVax Day 1 does not have to coincide with Pembrolizumab dosing
  Interventions: Radiation: Radiation Therapy; Biological: Personalized NeoAntigen Peptides; Drug: Pembrolizumab; Biological: Poly-ICLC
- Coh 1d: Std RT+TMZ Followed by 6 Cyc TMZ + NeoVax + Pembro (Experimental): • RT: Standard RT (60Gy) + concurrent daily temozolomide (TMZ) over 6 weeks. Concurrent TMZ @ 75 mg/m2/day for 6 weeks.
  Followed by:
  * 6 cycles of Adjuvant temozolomide (TMZ): Starts 4-6 weeks after completion of RT. TMZ (150-200 mg/m2/day) on days 1-5 of each 28-day cycle for 6 cycles.
  * Pembrolizumab: Starts 1-4 weeks after completion of NeoVax priming, and continues every 3 weeks for up to 2 years
  * NeoVax: Starts in the Adjuvant setting - as soon as available after RT - and is administered on days 1, 4, 8, 15, 22 [priming doses], 78 and 134 [booster doses] o NeoVax Day 1 does not have to coincide with Pembrolizumab dosing
  Interventions: Radiation: Radiation Therapy; Biological: Personalized NeoAntigen Peptides; Drug: Pembrolizumab; Drug: Temozolomide; Biological: Poly-ICLC

INTERVENTIONS:
Radiation: Radiation Therapy — Standard radiotherapy (approximately 60 Gy over 6 weeks)
  Other Names: RT, XRT
Biological: Personalized NeoAntigen Peptides — NeoVax Vaccine (Personalized NeoAntigen Peptides + Poly-ICLC) will be administered on an individual basis using a dosing schedule that incorporates both priming and boost phases.
Drug: Pembrolizumab — Pembrolizumab will be administered every 3 weeks at a flat dose of 200 mg intravenously. Pembrolizumab should be administered as a 30 minute IV infusion (Pembrolizumab treatment cycle intervals may be increased due to toxicity per protocol).
  Other Names: MK-3475, Keytruda
  Arms: Coh 1a: Pembrolizumab w Std RT Followed by NeoVax + Pembro; Coh 1b: Std RT Followed by NeoVax + Pembrolizumab; Coh 1c: Std RT (+ 1 dose Pembro) Followed by NeoVax & Pembo; Coh 1d: Std RT+TMZ Followed by 6 Cyc TMZ + NeoVax + Pembro
Drug: Temozolomide — Concurrent Temozolomide (TMZ) = 75 mg/m2/day for 6 weeks, administered with XRT
  Other Names: Concurrent temozolomide; Concurrent TMZ
  Arms: Coh 1d: Std RT+TMZ Followed by 6 Cyc TMZ + NeoVax + Pembro
Drug: Temozolomide — Adjuvant Temozolomide (TMZ) = 150 mg/m2/day on days 1-5 of each 28-day cycle for up to 6 adjuvant cycles
  Other Names: Adjuvant temozolomide; Adjuvant TMZ
  Arms: Coh 1d: Std RT+TMZ Followed by 6 Cyc TMZ + NeoVax + Pembro
Biological: Poly-ICLC — NeoVax Vaccine (Personalized NeoAntigen Peptides + Poly-ICLC) will be administered on an individual basis using a dosing schedule that incorporates both priming and boost phases.
  Other Names: Hiltonol

SUMMARY:
This research study is studying a new type of vaccine as a possible treatment for patients with glioblastoma. This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the intervention to use for further studies. "Investigational" means that the intervention is being studied and that research doctors are trying to find more about it. It also means that the FDA (U.S. Food and Drug Administration) has not approved the Personalized NeoAntigen Cancer Vaccine for any use in patients, including people with glioblastoma.

The purpose of the initial study cohort (Cohort 1) is to determine if it is possible to make and administer safely a vaccine against glioblastoma by using information gained from specific characteristics of the participants tumor. It is known that glioblastomas have mutations (changes in genetic material) that are specific to an individual patient's tumor. These mutations can cause the tumor cells to produce proteins that appear very different from the body's own cells. It is possible that these proteins used in a vaccine may induce strong immune responses, which may help the body fight any tumor cells that could cause the glioblastoma to come back in the future.

Three additional cohorts (1a, 1b, & 1c) were added to the study following completion of accrual to the original study cohort (cohort 1). Each new cohort receives NeoVax and radiation therapy as administered to cohort 1 and will also receive pembrolizumab: cohort 1a patients will start pembrolizumab w/in 2 weeks after start of RT, and continue every 3 weeks for up to 2 years; cohort 1b patients will start pembrolizumab 2-4 weeks after completion of NeoVax priming, and continue every 3 weeks for up to 2 years; cohort 1c patients will receive a single dose of pembrolizumab administered within 2 weeks after start of RT, re-start 2-4 weeks after completion of NeoVax priming, and continue every 3 weeks for up to 2 years. The rationale for adding these new cohorts is: 1) to assess the safety and feasibility of NeoVax when administered with pembrolizumab; and 2) to determine if the timing of anti-PD-1 administration impacts the immunogenicity of NeoVax.

An additional sub-study cohort (1d) is being added for patients whose tumor is MGMT-methylated. Cohort 1d will enroll patients with tumors for which the MGMT status is methylated or partially methylated; patients on cohort 1d will receive standard daily temozolomide during radiation and as adjuvant therapy for up to six cycles following completion of radiation therapy. The rationale for adding cohort 1d is to determine the safety and feasibility of NeoVax when administered with pembrolizumab and temozolomide.

DETAILED DESCRIPTION:
It is known that glioblastomas have mutations that are specific to an individual patient's tumor. These mutations can cause the tumor cells to produce proteins that appear very different from the body's own cells. It is possible that these proteins used in a vaccine may induce strong immune responses, which may help the body fight any tumor cells that could cause glioblastoma to recur.

Methylguanine methyltransferase (MGMT) is a DNA repair protein which can be increased in some cancers, including glioblastoma. MGMT works to repair the DNA of cancer cells that are damaged by treatment. If a tumor is found to be "unmethylated", it means there is more MGMT present in the tumor than one that is "methylated".

Methylation of MGMT is believed to make tumor cells more responsive to drugs like temozolomide. Studies have shown that temozolomide provides a very small improvement in outcome for many patients whose glioblastoma is MGMT-unmethylated.

Patients with glioblastoma usually receive six weeks of radiation with a daily chemotherapy called temozolomide after their surgery, followed by six to twelve months of additional temozolomide. In this study, only participants whose tumors are MGMT-methylated will receive temozolomide; those participants whose tumors are MGMT-unmethylated will not receive temozolomide, as studies have shown that temozolomide provides a very small improvement in outcome for many patients whose glioblastoma is MGMT-unmethylated.

On this trial, an initial cohort of participants (Cohort 1) will receive the Personalized NeoAntigen Vaccine (5 priming doses and 2 booster doses over ~ 20 weeks) after having completed six weeks of standard radiation. The study will examine the safety of the vaccine when given at several different time points and will examine the participant blood cells for signs that the vaccine induced an immune response.

Three additional cohorts (1a, 1b, & 1c) were added to the study following completion of accrual to the original study cohort (cohort 1). Each new cohort receives NeoVax and radiation therapy as administered to cohort 1 and will also receive pembrolizumab: cohort 1a patients will start pembrolizumab w/in 2 weeks after start of RT, and continue every 3 weeks for up to 2 years; cohort 1b patients will start pembrolizumab 2-4 weeks after completion of NeoVax priming, and continue every 3 weeks for up to 2 years; cohort 1c patients will receive a single dose of pembrolizumab administered within 2 weeks after start of RT, re-start 2-4 weeks after completion of NeoVax priming, and continue every 3 weeks for up to 2 years.

The rationale for adding cohorts 1a, 1b and 1c is: 1) to assess the safety and feasibility of NeoVax when administered with pembrolizumab; and 2) to determine if the timing of anti-PD-1 administration impacts the immunogenicity of NeoVax.

An additional sub-study cohort (1d) is being added for patients whose tumor is MGMT-methylated. Cohort 1d will enroll patients with tumors for which the MGMT status is methylated or partially methylated; patients on cohort 1d will receive standard daily temozolomide during radiation and as adjuvant therapy for up to six cycles following completion of radiation therapy. The rationale for adding cohort 1d is to determine the safety and feasibility of NeoVax when administered with pembrolizumab and temozolomide.

ELIGIBILITY:
I. Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study (labs/tests/assessments within 14 days prior to initial study registration unless otherwise specified)

* Participant is willing and able to give written informed consent
* Pathologically confirmed WHO grade IV glioblastoma or variants (gliosarcoma, glioblastoma with oligodendroglial features, giant cell glioblastoma) with adequate tumor material for genomic sequencing. Participants will be eligible if the original diagnosis was a lower grade glioma and a subsequent histologic diagnosis of glioblastoma or its variants was made, and patient received no prior therapy other than surgery

  * Patients with a diagnosis of astrocytoma with molecular features of glioblastoma will be considered eligible for trial.
  * In addition, patients with IDH-mutated tumors will also continue to be eligible for trial, despite the release of updated WHO disease classifications in 2021.
* The tumor must be primarily supratentorial in location as determined by diagnostic imaging performed preoperatively
* Radiographic contrast enhancement attributable to residual tumor on post-operative imaging performed within 72 hours of resection must not exceed 1 cm in maximal diameter in biperpendicular plances (greater than 1 cm in one plane but less than 1 cm in other planes will be allowed)
* CT or MRI within 14 days prior to start of study therapy (NOTE: This criterion does not apply to Cohort 1d participants who are registering after having initiated standard of care therapy.)
* Age ≥18 years
* Karnofsky performance status ≥ 70
* Participant is a candidate for, and agrees to receive conventional external beam radiotherapy. (Patients screening for Cohort 1d can be actively receiving - or already completed - their first line conventional external beam radiotherapy.)
* No corticosteroid dosing within 5 days of radiation therapy initiation (Cohorts 1a, 1b, 1c, & 1d).
* Normal hematologic, renal and hepatic function as defined below:

  * ANC: greater or equal to 1,000 /mcl
  * Platelets: greater than or equal to 100,000 /mcl
  * Hemoglobin: greater than or equal to 9 gm/dl or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
  * International normalized ratio (INR) or prothrombin time: less than or equal to 1.5 times institutional ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated partial thromboplatin time (aPTT): less than or equal to 1.5 X institutional ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Serum creatinine: less than or equal to 1.5 X institutional ULN OR Measured or calculated creatinine clearance ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
  * Total bilirubin: less than or equal to 1.5 X institutional ULN (or less than or equal to 3.0 X institutional ULN for Gilbert's Syndrome) OR Direct bilirubin ≤ institutional ULN for subjects with total bilirubin levels > 1.5 institutional ULN
  * AST (SGOT) and ALT (SGPT): less than or equal to 2.5 X institutional ULN (or less than or equal to 5.0 X institutional ULN for Gilbert's Syndrome)
* MGMT promoter methylation status determined by an institutional CLIA-approved laboratory using a methylation specific PCR assay
* Adequate tumor content as determined by institutional pathologist for nucleic acid extraction and DNA sequence analysis
* Patients unable to undergo magnetic resonance (MR) imaging because of non-compatible devices can be enrolled, provided CT scans are obtained and are of sufficient quality. Patients without non-compatible devices may not have CT scans performed to meet this requirement
* An interval of at least 3 weeks between prior surgical resection to start of study therapy (or one week for stereotactic biopsy to start of study treatment);
* Women of childbearing potential (WOCBP) must have a negative pregnancy test (minimum sensitivity 25 IU/L or equivalent of HCG) before entry onto the trial, because the effects NeoVax on the developing human fetus are unknown
* Participants cannot be breast feeding;
* Female participants enrolled in the study, who are not free from menses for greater than or equal to 2 years, post hysterectomy/oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from sexual activity throughout the study, starting with visit 1 through 120 days after the last dose of the study therapy;
* Approved contraceptive methods include for example; intra uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception;
* Male participants must agree to use an adequate method of contraception starting with the first dose of radiation therapy through 120 days after the last dose of study therapy.

II. Exclusion Criteria:

Participants who exhibit any of the following conditions at either screening timepoint will not be eligible for admission into or continuation on the study

* Stereotactic biopsy (without further resection);
* Tumor primarily localized in the infratentorial compartment or spinal cord - tumors with limited infratentorial compartment or spinal cord involvement are eligible;
* Radiographic or cytologic evidence of diffuse leptomeningeal extension - tumors with limited subependymal involvement are eligible;
* Participants who have received or plan to receive any additional treatment for glioblastoma aside from surgical resection and conventional radiotherapy (Cohort 1) and pembrolizumab (cohorts 1a, 1b and 1c) and temozolomide (cohort 1d), including - but not limited to - temozolomide (cohorts 1, 1a, 1b and 1c), stereotactic radiosurgery, placement of Gliadel (carmustine; BCNU) wafers, any other intratumoral or intracavitary treatment, brachytherapy, Novo-Tumor Treating Fields (Optune), or investigational therapeutic agents. (Cohort 1d participants may have already initiated or completed their RT with concomitant TMZ, and may have initiated their adjuvant TMZ at the time of study entry as long as they do not have evidence of progressive disease and have undergone a leukopheresis or blood draw with adequate mononuclear cell collection.)
* Concomitant therapy with any anti-cancer agents, other investigational anti-cancer therapies, or immunosuppressive agents including but not limited to methotrexate, chloroquine, azathioprine, etc. within six months of study participation;
* History of severe allergic reactions attributed to any vaccine therapy for the prevention of infectious diseases;
* Active, known, or suspected autoimmune disease or immunosuppressive conditions that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs) with the exception of vitiligo, type 1 diabetes, residual autoimmune-related hypothyroidism requiring hormone replacement, or psoriasis not requiring systemic treatment. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known chronic infections with HIV, hepatitis B (HBV) or C (HCV), Hepatitis B virus DNA and testing for HCV RNA must be undetectable.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring treatment, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia;
* Any underlying medical condition, psychiatric condition or social situation that in the opinion of the investigator would compromise study administration as per protocol or compromise the assessment of AEs;
* Planned major surgery;
* Pregnant women are excluded from this study because personalized neoantigen peptides and poly-ICLC are agents with unknown risks to the developing fetus. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with personalized neoantigen peptides and poly-ICLC, nursing women are excluded from this study;
* Individuals with a history of an invasive malignancy are ineligible except for the following circumstances; a) individuals with a history of invasive malignancy are eligible if disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; b) individuals with the following cancers are eligible if diagnosed and treated - carcinoma in situ of the breast, oral cavity or cervix and basal cell or squamous cell carcinoma of the skin;

Coh 1a/1b/1c/1d Exclusions:

* Hypersensitivity to pembrolizumab or any of its excipients.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used investigational device within 4 weeks of the first dose of treatment. (NOTE: Participation in a clinical trial evaluating interventions for purposes other than GBM therapy is not a basis for exclusion, and may be permitted pending prospective approval of Principal Investigator or designee.)
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., less than or equal to Grade1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., less than or equal to Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with less than or equal to Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, subject must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
  * Note: Cohort 1d participants may have already received their radiation therapy with concomitant temozolomide, and may have initiated their adjuvant temozolomide, at the time of study entry as long as they do not have evidence of progressive disease and have undergone a leukopheresis or blood draw with adequate mononuclear cell collection.
* Has a known history of active TB (Bacillus Tuberculosis)
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate proved the disease is stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability;
* Has known history of non-infectious pneumonitis/ interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has received a live vaccine within 30 days of planned start of study therapy. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and Typhoid vaccine.

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Cohorts 1, 1a, 1b, & 1c: Number of participants with Adverse Events as a measure of safety and tolerability | 2 Years
  To evaluate the safety and tolerability of administering NeoVax plus pembrolizumab among newly diagnosed glioblastoma patients with MGMT unmethylated tumors
Cohorts 1d: Number of participants with Adverse Events as a measure of safety and tolerability | 2 Years
  To evaluate the safety and tolerability of administering NeoVax plus pembrolizumab and temozolomide among newly diagnosed glioblastoma patients with MGMT methylated/partially methylated tumors
Cohort 1: Number of participants with at least 10 actionable peptides as a measure of study feasibility | 2 Years
  This information will be used to determine the feasibility of generating and administering NeoVax in participants with newly diagnosed glioblastoma.
Cohort 1: Number of participants who are clinically able to initiate post-RT vaccine therapy within 12 weeks or less from date of surgery | 2 Years
  This information will be used to determine the feasibility of generating and administering NeoVax in participants with newly diagnosed glioblastoma.

SECONDARY OUTCOMES:
All Cohorts: Number of participants who achieve IFN-γ T-cell response at week 16 via ELISPOT assessments | 2 Years
  This information will be used to assess the induction of neoantigen-specific cellular immune responses following administration of Neovax with or without pembrolizumab.
Cohorts 1, 1a, 1b, & 1c: Number of participants who are alive without progression at eight months after surgery resection | 2 Years
  Estimate of the proportion of participants alive without disease progression at eight months after resection.
Cohort 1d: Number of participants who are alive without progression at 11 months after surgery resection | 2 years
  Estimate of the proportion of participants alive without disease progression at eleven months after resection.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts